Ministry of Higher Education and Scientific Research Al-Nahrain University High Institute for Infertility Diagnosis and Assisted Reproductive Technologies





## Study the Effects of Intrauterine flushing with Low Dose Human Chorionic Gonadotrophin on Endometrial Receptivity and ICSI Outcome



OCTOBER 16, 2024

CHAPTER FOUR RESULTS

## Statistical analysis

The data analyzed using Statistical Package for Social Sciences (SPSS) version 26. The data presented as mean, standard deviation and ranges. Categorical data presented by frequencies and percentages. Independent t-test and Analysis of Variance (ANOVA) (two tailed) was used to compare the continuous variables accordingly. Paired t-test was used to compare the continuous variables on pickup day and on transfer day. Chi square test was used to assess the association between categorical variables, while fisher exact test was used instead when the expected frequency was less than 5. A level of P – value less than 0.05 was considered significant.